CLINICAL TRIAL: NCT01353833
Title: Dose-effect Relationship of Repeated Administration of Low-dose IL-2 Versus Placebo on the Kinetic of Regulatory T Cells in Patients With Type 1 Diabetes
Brief Title: Dose-effect Relationship of Low-dose IL-2 in Type 1 Diabetes
Acronym: DF-IL2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P101101; 2010-024499-24 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2011-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IL2-4 (Placebo Comparator)
  Interventions: Drug: Aldesleukin
- IL2-2 (Experimental): 1 millions IU of IL-2 per day
  Interventions: Drug: Aldesleukin
- IL2-3 (Experimental): 3 millions IU of IL-2 per day
  Interventions: Drug: Aldesleukin
- IL2-1 (Experimental): 0.33 millions IU of IL-2 per day
  Interventions: Drug: Aldesleukin

INTERVENTIONS:
Drug: Aldesleukin — 0.33 ; 1 ; 3 ; 0 millions IU of IL-2 per day for arm 1 to 4, respectively. 1 s.c. injection per day for 5 days.
  Other Names: IL2

SUMMARY:
IL-2 is an inducer of regulatory T cells (Treg), a population of lymphocytes that fail to control the autoimmune destruction of beta-cells in patients with Type 1 Diabetes (T1D). The investigators recently showed that low dose IL-2 is well tolerated in patients with an autoimmune disease. The investigators aim to use IL-2 to induce/stimulate Treg in T1D patients. This study will investigate the dose effect relationship of low dose IL-2 for Treg induction such as to optimize the risk benefit ratio for this treatment in T1D. By Treg induction, the investigators aim to protect the remaining/regenerating β-cells from autoimmune destruction, thus improving or even curing T1D.

DETAILED DESCRIPTION:
Rationale:

Type 1 diabetes (T1D) results from an autoimmune destruction of beta-pancreatic cells that regulatory T cells (Treg) fail to control. This is in part due to a deficit in production of, or response to, interleukin 2 (IL-2). This cytokine is essential to Treg development, survival and function. Importantly, while IL-2 also contributes to the activation of effector T cells (Teff), IL-2/IL-2 receptor signal transduction threshold is much lower for Treg than Teff. Thus low-dose IL-2 could be a specific Treg inducer/stimulator.

The investigators then recently showed that low-dose IL-2 could cure recent onset diabetes in NOD mice that develop spontaneous diabetes considered as the best model of human T1D. A 5-day treatment with IL-2 could cure over 30% of the mice versus 0% for controls.

With these premises, the investigators propose to explore if Treg induction could be obtained in patients who may have a deficit in production of, or response to, IL-2. Defining the dose effect relationship of low dose IL-2 for Treg induction will optimize the risk benefit ratio for IL-2 in T1D.

Principal objective:

To define the dose-effect relationship of low dose IL-2 for Treg induction in patient with recent onset diabetes

Evaluation Criteria:

* Efficacy Kinetic variation of Treg proportions within CD4+ T cells in peripheral blood from Day+0 to Day+60.
* Tolerance Evaluation by clinical exams, laboratory tests and monitoring of side effects. The criterion for terminating the study will be the occurrence of one serious unexpected side effect in the month following IL-2 first administration in at least 2 patients.

Study plan:

After inclusion (Day0), the patient receives a 5-day course of IL-2 or placebo. Patients are randomized in 4 arms receiving either a placebo, or IL-2 doses of 0,33 - 1 or 3 millions UI/day. Laboratory follow-up of peripheral blood T cell subsets will be performed at D0 to D6 (daily), D15, D22 and D60 by immunophenotyping and transcriptomics.

Tolerance will be evaluated at D0-6, D15, D22 and D60.

Methodology:

Double blind placebo controlled randomized study, with 4 parallel groups. Patients will have T1D of autoimmune origin attested by the presence of auto-antibodies (at least one of: anti-islet, anti-GAD, anti-IA2 or anti-ZnT8), with a diagnostic inferior or equal to 24 months.

Study length:

Study length = 9 months Patient participation = 2 months Inclusion period = 6 months

ELIGIBILITY:
Inclusion Criteria:

* Age [18-50] years;
* With a T1D:
* Treated with insulin for ≤ 2 years,
* With at least one auto-antibody among: anti-islet, anti-GAD, anti-IA2, anti-ZnT8 ;
* No clinically relevant abnormal value for hematology, biochemistry, liver and kidney function
* Lymphocyte [1000-4000]/ mm3
* Informed consent signed by the patient and the investigator before any intervention necessary for the trial.

Exclusion Criteria:

* Contra-indications to IL2 :
* Hypersensibility to IL-2 or its excipients,
* Severe cardiopathy
* Ongoing infection requiring antibiotherapy,
* O2 Saturation ≤ 90 %
* Severe impairment of a vital organ
* Previous organ allograft
* Non authorized concomitant treatment : i.e. immuno-modulators, cytotoxic, drug modifying glycemia
* Cancer progressing or cured for less than 5 years except for primary basal cell carcinoma or carcinoma in situ of the uterine cervix.
* Participation to another clinical investigation in < 3 months
* Pregnant or lactating women
* Male or female in age of procreation without efficient contraception during the study
* No affiliation to National Health Insurance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Kinetic parameters of Treg proportions variation within CD4+ T cells in peripheral blood | from Day+0 to Day+60

SECONDARY OUTCOMES:
Improvement of residual secretion of insulin assessed by the AUC of peptide C during a standardized test meal in IL-2 vs placebo treated patients | at Day+0 and Day+60

CONTACTS AND LOCATIONS:
Overall Officials: Davis Klatzmann, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Hartemann A, Bensimon G, Payan CA, Jacqueminet S, Bourron O, Nicolas N, Fonfrede M, Rosenzwajg M, Bernard C, Klatzmann D. Low-dose interleukin 2 in patients with type 1 diabetes: a phase 1/2 randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):295-305. doi: 10.1016/S2213-8587(13)70113-X. Epub 2013 Oct 8. PMID 24622415